CLINICAL TRIAL: NCT04726891
Title: Feasibility of the First Known Adaptive Intervention Delivering Innovative Exercise Program Optimized for People With SCI
Brief Title: Feasibility of the First Known Adaptive Intervention for People With SCI
Acronym: SMART-HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, Jereme Wilroy, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 645335; 645335 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injuries
Keywords: exercise; behavioral coaching
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: sequential multiple assignment randomized trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Continued M2M + SNS for 9 weeks (Active Comparator): Participants who successfully watch and exercise at or above 40 minutes per week will continue doing M2M + SNS for the remaining 9 weeks of the study.
  Interventions: Behavioral: Movement-2-Music + Social Networking Support
- Augmented M2M + SNS + IBC for 9 weeks (Active Comparator): Some participants with sub-optimal adherence in the first treatment stage will be randomized to one of two treatment groups in the second treatment stage. these participants will receive M2M plus social networking support augmented with individualized behavioral coaching. Individualized behavioral coaching involves a weekly coaching session to improve self-regulatory skills based on prior and individualized exercise prescription. The exercise prescriptions are determined by the coach and individual based on their current activity level and a 4-week goal. An example of tailoring the exercise prescribed involves setting a goal of completing the exercise routine one time for the upcoming week instead of three times. The coach will be trained in motivational interviewing to help the participant modify their exercise habits.
  Interventions: Behavioral: Movement-2-Music + Social Networking Support
- Switched M2M Live for 9 weeks (Active Comparator): The remaining half of participants with sub-optimal adherence in the first treatment stage will switch to another M2M-based home exercise intervention, M2M Live. M2M Live involves one-on-one tele-exercise training with an M2M instructor, which provides accountability and immediate, tailored feedback along with custom movements and music. During the first week of M2M Live, the participant will set a schedule to meet with the M2M instructor 1 time each week for an exercise session. The M2M Live instructors are also trained in motivational interviewing in order to coach participants through any barriers to changing their exercise behavior.
  Interventions: Behavioral: Movement-2-Music + Social Networking Support
- Continued M2M + IBC for 6 weeks (Active Comparator): Participants who successfully watch and exercise at or above 40 minutes per week will continue doing M2M + SNS for the remaining 6 weeks of the study.
  Interventions: Behavioral: Movement-2-Music + Social Networking Support
- Augmented M2M + SNS + IBC for 6 weeks (Active Comparator): Some participants with sub-optimal adherence in the first treatment stage will be randomized to one of two treatment groups in the second treatment stage. these participants will receive M2M plus social networking support augmented with individualized behavioral coaching. Individualized behavioral coaching involves a weekly coaching session to improve self-regulatory skills based on prior and individualized exercise prescription. The exercise prescriptions are determined by the coach and individual based on their current activity level and a 4-week goal. An example of tailoring the exercise prescribed involves setting a goal of completing the exercise routine one time for the upcoming week instead of three times. The coach will be trained in motivational interviewing to help the participant modify their exercise habits.
  Interventions: Behavioral: Movement-2-Music + Social Networking Support
- Switched M2M Live for 6 weeks (Active Comparator): The remaining half of participants with sub-optimal adherence in the first treatment stage will switch to another M2M-based home exercise intervention, M2M Live. M2M Live involves one-on-one tele-exercise training with an M2M instructor, which provides accountability and immediate, tailored feedback along with custom movements and music. During the first week of M2M Live, the participant will set a schedule to meet with the M2M instructor 1 time each week for an exercise session. The M2M Live instructors are also trained in motivational interviewing in order to coach participants through any barriers to changing their exercise behavior.
  Interventions: Behavioral: Movement-2-Music + Social Networking Support

INTERVENTIONS:
Behavioral: Movement-2-Music + Social Networking Support — The primary goal of the proposed research is to conduct a 12-week pilot study of the SMART-HEALTH intervention in 30 individuals with SCI. There are several unique features of this study design, including a novel adapted exercise program (M2M), instructor-led, individualized training (M2M Live; described in D.2.1), individualized behavioral coaching, and social networking support.
  Other Names: Individual Behavioral Coaching; Movement-2-Music Live

SUMMARY:
The overall goal of the proposed research is to conduct a pilot study to test the feasibility and acceptability of a home-based exercise intervention (SMART-HEALTH). The primary purpose of the pilot study is to assess the feasibility of intervention delivery (Aim 1), the acceptability of the intervention by participants (Aim 2) and estimate effect sizes for a future trial (Aim 3).

DETAILED DESCRIPTION:
The proposed project aims to address low adherence to exercise interventions among people with SCI. Specifically, we will conduct a 12-week pilot study of a SMART design using a telehealth-delivered intervention previously developed for people with mobility disability as the primary intervention strategy. This intervention, Movement-to-Music (M2M), has been previously packaged as a collection of videos disseminated through an app on a weekly schedule. M2M has been shown to effectively improve physiological outcomes among people with a neurological disability, including SCI. Data collection will include accelerometer-based measurement of physical activity and sleep during the intervention, a 3-day physical activity recall, and assessment of physiological (e.g., grip strength) and psychosocial factors (i.e., depression, anxiety) collected before and after intervention. Social Cognitive Theory has been used successfully in past studies to improve many health behaviors. Thus, it will be utilized into SMART-HEALTH as the following constructs: self-efficacy, self-regulation, social support, and outcome expectations.

A sample of individuals with SCI will be randomized to 3 weeks or 6 weeks of M2M with social networking support for the first treatment stage. Depending on adherence, they will either continue with the intervention received in the first treatment stage or be randomized a second time. Specifically, participants with high adherence (40 or more minutes) will continue M2M with social networking support, while those with low adherence (less than 40 minutes) will be randomized to an augmented arm that includes individualized behavioral coaching or to an arm that switches to M2M Live. The second treatment stage will last until the participant has completed a total of 12 weeks on the program. The social networking support, individualized behavioral coaching, and M2M Live sessions will be completed through secure videoconferencing on the mobile health platform, which will allow a singular location for tracking intervention activity. All security features of the integrated videoconferencing software will be used, including passwords and waiting rooms.

M2M. In the first treatment stage, all participants will receive M2M as the evidence-based home exercise intervention. M2M is provided in the form of an exercise routine that includes aerobic and strength training set to music. Each week the participants will receive a set of exercise videos, which they will be asked to complete 3 times during the week. Exercise videos begin with a low dose of minutes, approximately 10 to 15 minutes for a total of 40 minutes for the week, and increase by 3-5 minutes each week.

Social Networking Support. In the first treatment stage, all participants will also receive social networking support. The group will also be able to communicate through the mobile health platform via features such as messaging, posting, commenting, and liking. Each week a discussion board will provide an opportunity for participants to post comments concerning the week's exercise content, weekly article, and/or their experience with the program that week.

Individual Behavioral Coaching. Some participants with sub-optimal adherence in the first treatment stage will be randomized to one of two treatment groups in the second treatment stage. Half of these participants will receive M2M plus social networking support augmented with individualized behavioral coaching.

M2M Live. The remaining half of participants with sub-optimal adherence in the first treatment stage will switch to another M2M-based home exercise intervention, M2M Live. This involves one-on-one tele-exercise training with an M2M instructor. During the first week of M2M Live, the participant will set a schedule to meet with the M2M instructor one time per week for an exercise session. The exercise session will be recorded and posted for the participant to complete 2 additional times.

ELIGIBILITY:
Inclusion Criteria:

* SCI greater than or equal to 1 year after injury
* Wheelchair User
* Able to use arms for exercise
* 18+ years old
* Sedentary (<60 minutes of exercise/week)

Exclusion Criteria:

* Cognitive Impairment (Folstein's Mini-Mental State Exam Score < 24)
* Depression (Centers for Epidemiological Studies Depression Scale Score > 16)
* Poorly controlled blood pressure (SBP > 159 or DBP > 95 mmHg)
* Cardiovascular disease event within the past 6 months, severe pulmonary disease, kidney failure
* Active pressure ulcers

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Physical Activity | baseline, 4-weeks, 8-weeks, and 12 weeks
  Physical Activity Recall Among people with Spinal Cord Injury (PARA-SCI) Instrument will be used to assess minutes of physical activity. Designed to estimate 3-day summary values for physical activity, including intensity (mild, moderate, or vigorous), duration, and modality (aerobic or strength training), which results in providing total minutes of moderate to vigorous physical activity. The higher number of minutes the better.

SECONDARY OUTCOMES:
Strength | baseline and 12 weeks
  Grip strength
Respiratory functioning | baseline and 12 weeks
  Peak Expiratory Volume measured by spirometer
Blood pressure | baseline and 12 weeks
  Two readings prior to exercise using digital blood pressure cuff.
Heart rate | baseline and 12 weeks
  Two readings prior to exercise using digital blood pressure cuff.
Physical activity self-efficacy scale | baseline and 12 weeks
  Survey of social cognitive theory construct.
Outcomes expectations for exercise scale | baseline and 12 weeks
  Survey of social cognitive theory construct.
demographics | baseline and 12 weeks
  questionnaire including age, sex, race, ethnicity
sleep disturbance | baseline and 12 weeks
  Secondary health conditions NIH PROMIS
Depression | baseline and 12 weeks
  Secondary health conditions NIH PROMIS
Pain intensity | baseline and 12 weeks
  Secondary health conditions NIH PROMIS
Anxiety | baseline and 12 weeks
  Secondary health conditions NIH PROMIS

CONTACTS AND LOCATIONS:
Overall Officials: Jereme D Wilroy, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Lakeshore Foundation, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilroy J, Kim Y, Lai B, Young HJ, Giannone J, Powell D, Thirumalai M, Mehta T, Rimmer J. Increasing Physical Activity in Persons With Spinal Cord Injury With an eHealth-Based Adaptive Exercise Intervention: Protocol for a Sequential Multiple Assignment Randomized Trial. JMIR Res Protoc. 2023 Jul 27;12:e47665. doi: 10.2196/47665. PMID 37498650